CLINICAL TRIAL: NCT00976625
Title: Persistent Diastolic Dysfunction Late After Valve Replacement in Severe Aortic Regurgitation
Brief Title: Diastolic Dysfunction in Aortic Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: University Hospital Bern, Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-32 16.9.1992 (Zürich)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Aortic Regurgitation
Keywords: diastolic function; aortic regurgitation; aortic valve replacement; left ventricular hypertrophy; myocardial structure; LV remodeling; Muscular regression; LV fibrous tissue
MeSH Terms: conditions — Aortic Valve Insufficiency; Hypertrophy, Left Ventricular | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control group without intervention. Treatment group with aortic valve replacement.
- 2 (Other)
  Interventions: Procedure: Aortic Valve Replacement

INTERVENTIONS:
Procedure: Aortic Valve Replacement — Surgical valve replacement of the aorta
  Arms: 2

SUMMARY:
Follow-up study in patients with severe aortic regurgitation after successful valve replacement. Systolic and diastolic function were assessed and persistent diastolic dysfunction was observed late (7-10 years) after operation.

DETAILED DESCRIPTION:
Background

Patients with severe aortic regurgitation show eccentric LV hypertrophy and structural changes of the myocardium. Reversibility of functional and structural changes after successful valve replacement may be limited. Persistent diastolic dysfunction has been observed in the present study late after aortic valve replacement. This finding has been explained by incomplete regression of the extra-cellular matrix 7 years after valve replacement. Interstitial fibrosis remains unchanged compared to the preoperative situation but was increased early after operation due to the reduction in LV muscle mass. Regression of LV hypertrophy was 40% after 2 and 55% after 7 years of valve replacement. Myocardial muscle fibers decreased slightly but remained hypertrophied even late after operation. Interstitital fibrosis was found to be positively correlated to myocardial stiffness and inversely to LV ejection fraction.

Thus, persistent diastolic dysfunction with maintained systolic ejection performance can be observed late after successful valve replacement in patients with severe aortic regurgitation. Altered diastolic function has been associated with increased filling pressures during strenuous exercise with signs of dyspnea.

Objective

Evaluation of myocardial structure and function in patients with chronic volume overload before and after valve replacement(LV-remodeling).

Methods

Pressure-volume measurements and myocardial biopsy samples for assessing myocardial function and structure.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic regurgitation
* Successful valve replacement
* Informed consent
* Sinus rhythm
* No comorbidities
* No bundle branch block
* No pregnancy

Exclusion Criteria

* Unwillingness to undergo postop. cath
* diabetes mellitus
* arterial hypertension
* bleeding disorder
* pulmonary hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1996-01; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cardiac function and structure | 7-10 years

SECONDARY OUTCOMES:
LV hypertrophy and passive elastic properties | 7-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hess, Principal Investigator — University of Bern
Locations (1):
- Division of Cardiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Villari B, Sossalla S, Ciampi Q, Petruzziello B, Turina J, Schneider J, Turina M, Hess OM. Persistent diastolic dysfunction late after valve replacement in severe aortic regurgitation. Circulation. 2009 Dec 8;120(23):2386-92. doi: 10.1161/CIRCULATIONAHA.108.812685. Epub 2009 Nov 23. PMID 19933939